CLINICAL TRIAL: NCT05398640
Title: Expanded Access Program of AMTAGVI That is Out of Specification for Commercial Release
Status: Available | Type: Expanded Access
Sponsor: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IOV-EAP 402
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Unresectable Melanoma; Metastatic Melanoma
Keywords: LN-144; Lifileucel; Adoptive Cell Therapy; Cell Therapy; Tumor Infiltrating Lymphocytes; TIL; Immunotherapy
MeSH Terms: conditions — Melanoma | interventions — lifileucel

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: OOS AMTAGVI — Patients will undergo preparative lymphodepleting chemotherapy. Infusion of lifileucel is then given and is followed by administration of IL-2.
  Other Names: LN-144; Lifileucel

SUMMARY:
The objective of this expanded access protocol is to provide access to Out Of Specification (OOS) AMTAGVI treatment to patients.

DETAILED DESCRIPTION:
This program provides access to OOS AMTAGVI (lifileucel) that does not meet commercial release criteria but does meet Iovance clinical trial release criteria. Patients will be followed for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for treatment with AMTAGVI per United States Prescribing Information (USPI)
2. Have an AMTAGVI product manufactured for commercial treatment; however, the final manufactured product did not meet commercial release criteria but was deemed safe and acceptable for release after risk/benefit assessment
3. Patients of childbearing potential or those with partners of childbearing potential must be willing to practice an approved method of highly effective birth control during treatment and for 12 months after receiving the last protocol-related therapy

Exclusion Criteria:

1. History of hypersensitivity to cyclophosphamide, mesna, fludarabine, or any component of lifileucel cryopreservation medium
2. Ongoing systemic infection
3. Cardiopulmonary or renal disorder which may make patient ineligible for treatment with cyclophosphamide, fludarabine or IL-2, at the discretion of the Treating Physician
4. Experience a significant worsening in clinical status that would, in the opinion of the Treating Physician, increase the risk of toxicities from treatment with lymphodepleting chemotherapy, AMTAGVI product that is out of specification, or IL-2
5. Any other condition, laboratory abnormality and/or pre-treatment assessment that places patient at unacceptable risk if they were to participate in the EAP based on the Treating Physician's judgment
6. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - HonorHealth, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - Stanford Hospital, Stanford, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Orlando Health Cancer Institute, Orlando, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Iowa Hospital, Iowa City, Iowa
  - The University of Kansas Cancer Center, Westwood, Kansas
  - University of Louisville - James Graham Brown Cancer Center, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University - Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - St. Lukes Hospital, Bethlehem, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center - U of Texas, Houston, Texas
  - Intermountain Healthcare, Salt Lake City, Utah
  - VCU Medical Center (Virginia Commonwealth University), Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin